CLINICAL TRIAL: NCT02829944
Title: Impact of Local Anesthetic Wound Infiltration on Postoperative Pain Following Cesarean Delivery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00069752
Record Dates: First submitted 2016-07-08; First posted 2016-07-12 (Estimated); Results first posted 2020-03-06 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-02

CONDITIONS: Pain
Keywords: Cesarean section
MeSH Terms: conditions — Pain | interventions — Ropivacaine; Ketorolac

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ropivacaine (Experimental): Subjects will receive 440 mg ropivacaine and 30 mg ketorolac. Infusion of study medication will start after the skin is sutured and will continue for 48 hours after cesarean delivery.
  Interventions: Drug: Ropivacaine; Drug: Ketorolac
- Placebo (Placebo Comparator): Subjects will receive saline placebo. Infusion of study medication will start after the skin is sutured and will continue for 48 hours after cesarean delivery.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ropivacaine
  Arms: Ropivacaine
Drug: Ketorolac
  Arms: Ropivacaine
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if the infusion of the local anesthetic ropivacaine (a numbing medicine) and the non-steroidal anti-inflammatory drug ketorolac (a pain killer similar to ibuprofen) through a catheter placed along the cesarean delivery incision, will reduce the pain experienced after cesarean section and need for narcotic pain medicine.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology (ASA) class 1,2, and 3
* English speaking women at a gestational age > 37 weeks
* scheduled for cesarean delivery under spinal or combined spinal epidural anesthesia

Exclusion Criteria:

* BMI > 50 kg/m2
* history of intravenous drug or opioid abuse
* previous history of chronic pain syndrome
* history of opioid use in the past week
* allergy or contraindication to any of the study medications
* non-English speaking

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf Habib, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States

REFERENCES:
- [Derived] Barney EZ, Pedro CD, Gamez BH, Fuller ME, Dominguez JE, Habib AS. Ropivacaine and Ketorolac Wound Infusion for Post-Cesarean Delivery Analgesia: A Randomized Controlled Trial. Obstet Gynecol. 2020 Feb;135(2):427-435. doi: 10.1097/AOG.0000000000003601. PMID 31923061

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study recruited participants from the Duke Labor and Delivery population, as they presented for scheduled Cesarean Delivery.
Groups:
- Placebo: Subjects will receive saline placebo. Infusion of study medication will start after the skin is sutured and will continue for 48 hours after cesarean delivery.
  Placebo
- Ropivacaine: Subjects will receive 440 mg ropivacaine and 30 mg ketorolac. Infusion of study medication will start after the skin is sutured and will continue for 48 hours after cesarean delivery.
  Ropivacaine
  Ketorolac
Period: Overall Study
Arm/Group | Placebo | Ropivacaine
Started | 44 | 40
Completed | 38 | 33
Not Completed | 6 | 7
Not completed — Physician Decision | 0 | 1
Not completed — Screen Failure | 2 | 2
Not completed — Inadequate Neuraxial Block | 1 | 1
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Catheter Displacement | 1 | 0
Not completed — Catheter broke | 0 | 1
Not completed — Staff unavailable | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Ropivacaine | Total
Number analyzed (Participants) | 38 | 33 | 71
Age, Continuous [Median (Inter-Quartile Range); unit: years]
  Age | 31.5 [27 to 36] | 30 [27 to 35] | 31 [27 to 36]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 33 | 71
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 37 | 31 | 68
  Not Hispanic or Latino | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 12 | 24
  White | 22 | 18 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 38 | 33 | 71

OUTCOME MEASURES:

1. Primary Outcome: Pain Score on Movement (Sitting in Bed From a Supine Position)
Description: Score reported on a scale of 0-10, with 0 being none and 10 being the worst imaginable
Time Frame: 24 hours after surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Placebo | Ropivacaine
Number analyzed (Participants) | 38 | 33
score on a scale | 5 [3 to 7] | 5 [4 to 6]

2. Secondary Outcome: Pain Scores at Rest
Description: Score reported on a scale of 0-10, with 0 being none and 10 being the worst imaginable
Time Frame: 2 hours
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Placebo | Ropivacaine
Number analyzed (Participants) | 38 | 33
score on a scale | 2 [0 to 3] | 0 [0 to 3]

3. Secondary Outcome: Pain Scores at Rest
Description: Score reported on a scale of 0-10, with 0 being none and 10 being the worst imaginable
Time Frame: 24 hours
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Placebo | Ropivacaine
Number analyzed (Participants) | 38 | 33
score on a scale | 2 [0 to 3] | 2 [0 to 3]

4. Secondary Outcome: Pain Scores at Rest
Description: Score reported on a scale of 0-10, with 0 being none and 10 being the worst imaginable
Time Frame: 48 hours
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Placebo | Ropivacaine
Number analyzed (Participants) | 38 | 33
score on a scale | 2 [1 to 4] | 2 [0 to 3]

5. Secondary Outcome: Opioid Consumption
Description: measured in mg oxycodone equivalents
Time Frame: 2 hours
Measure: Median (Inter-Quartile Range); unit: mg Oxycodone Equivalent
Arm/Group | Placebo | Ropivacaine
Number analyzed (Participants) | 38 | 33
mg Oxycodone Equivalent | 0 [0 to 0] | 0 [0 to 0]

6. Secondary Outcome: Opioid Consumption
Description: measured in mg oxycodone equivalents
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: mg Oxycodone Equivalent
Arm/Group | Placebo | Ropivacaine
Number analyzed (Participants) | 38 | 33
mg Oxycodone Equivalent | 5 [0 to 15] | 5 [0 to 15]

7. Secondary Outcome: Opioid Consumption
Description: measured in mg oxycodone equivalents
Time Frame: 48 hours
Measure: Mean (Inter-Quartile Range); unit: mg Oxycodone Equivalent
Arm/Group | Placebo | Ropivacaine
Number analyzed (Participants) | 38 | 33
mg Oxycodone Equivalent | 20 [10 to 35] | 10 [0 to 30]

8. Secondary Outcome: Time to First Rescue Analgesic
Time Frame: 48 hours
Measure: Mean (Inter-Quartile Range); unit: Minutes
Arm/Group | Placebo | Ropivacaine
Number analyzed (Participants) | 38 | 33
Minutes | 660 [99 to 1496] | 954 [244 to 1710]

9. Secondary Outcome: Number of Subjects Experiencing Nausea
Description: Asking patients whether or not they experienced the symptom in the preceding time-frame
Time Frame: 2 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ropivacaine
Number analyzed (Participants) | 38 | 33
Participants | 14 | 12

10. Secondary Outcome: Number of Subjects Experiencing Nausea
Description: Asking patients whether or not they experienced the symptom in the preceding time-frame
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ropivacaine
Number analyzed (Participants) | 38 | 33
Participants | 9 | 7

11. Secondary Outcome: Number of Subjects Experiencing Nausea
Description: Asking patients whether or not they experienced the symptom in the preceding time-frame
Time Frame: 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ropivacaine
Number analyzed (Participants) | 38 | 33
Participants | 4 | 1

12. Secondary Outcome: Number of Subjects Experiencing Vomiting
Description: Asking patients whether or not they experienced the symptom in the preceding time-frame
Time Frame: 2 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ropivacaine
Number analyzed (Participants) | 38 | 33
Participants | 7 | 8

13. Secondary Outcome: Number of Subjects Experiencing Vomiting
Description: Asking patients whether or not they experienced the symptom in the preceding time-frame
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ropivacaine
Number analyzed (Participants) | 38 | 33
Participants | 4 | 4

14. Secondary Outcome: Number of Subjects Experiencing Vomiting
Description: Asking patients whether or not they experienced the symptom in the preceding time-frame
Time Frame: 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ropivacaine
Number analyzed (Participants) | 38 | 33
Participants | 1 | 0

15. Secondary Outcome: Number of Subjects Experiencing Pruritus
Description: Score reported on a scale of 0-10, with 0 being none and 10 being the worst imaginable
Time Frame: 2 hours
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Placebo | Ropivacaine
Number analyzed (Participants) | 38 | 33
score on a scale | 4 [1 to 7] | 5.5 [3.5 to 8]

16. Secondary Outcome: Number of Subjects Experiencing Pruritus
Description: Score reported on a scale of 0-10, with 0 being none and 10 being the worst imaginable
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo | Ropivacaine
Number analyzed (Participants) | 38 | 33
units on a scale | 3.5 [0 to 7] | 4 [1 to 8]

17. Secondary Outcome: Number of Subjects Experiencing Pruritus
Description: Score reported on a scale of 0-10, with 0 being none and 10 being the worst imaginable
Time Frame: 48 hours
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Placebo | Ropivacaine
Number analyzed (Participants) | 38 | 33
score on a scale | 0 [0 to 0] | 0 [0 to 0]

18. Secondary Outcome: Patient Satisfaction With Postoperative Analgesia on a 0-10 Scale
Description: Score reported on a scale of 0-10, with 0 being not at all satisfied and 10 being completely satisfied
Time Frame: 48 hours
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Placebo | Ropivacaine
Number analyzed (Participants) | 38 | 33
score on a scale | 9.5 [8 to 10] | 8 [8 to 9.5]

19. Secondary Outcome: Number of Subjects With Chronic Pain
Description: Phone interview asking patient about presence of pain at incision site
Time Frame: 8 weeks
Population: Unable to make contact with 9 participants in the Placebo group and 13 participants in the Ropivacaine group.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ropivacaine
Number analyzed (Participants) | 29 | 20
Participants | 3 | 3

20. Secondary Outcome: Number of Subjects With Chronic Pain
Description: Phone interview asking patient about presence of pain at incision site
Time Frame: 6 months
Population: 28 participants in each group (Placebo and Ropivacaine) did not complete the interview.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ropivacaine
Number analyzed (Participants) | 10 | 5
Participants | 0 | 0

21. Secondary Outcome: Postpartum Depression, as Measured by the Edinburgh Postnatal Depression Scale
Description: Patients contacted over the phone completed screening with the EPDS, on a scale of 0-30. A score of over 13 indicate risk for postpartum depression
Time Frame: 8 weeks
Population: Unable to make contact with 9 participants in the Placebo group and 13 participants in the Ropivacaine group.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo | Ropivacaine
Number analyzed (Participants) | 29 | 20
units on a scale | 1 [0 to 4] | 0.5 [0 to 5]

22. Secondary Outcome: Postpartum Depression, as Measured by the Edinburgh Postnatal Depression Scale
Description: as for outcome 21
Time Frame: 6 months
Population: Unable to make contact with 19 participants in the Placebo group and 22 participants in the Ropivacaine group.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ropivacaine
Number analyzed (Participants) | 19 | 11
Participants | 3 | 1

23. Secondary Outcome: Pain Score on Movement
Description: Score reported on a scale of 0-10, with 0 being none and 10 being the worst imaginable
Time Frame: 48 hours after surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Placebo | Ropivacaine
Number analyzed (Participants) | 38 | 33
score on a scale | 5.5 [3 to 8] | 5 [4 to 6]

ADVERSE EVENTS:
Time Frame: From Anesthesia start to 48 hours postoperatively.
Description: Patients were asked at 2 hours, 24 hours and 48 hours to rate any symptoms on a scale of 0-10, with 0 being none at all and 10 being the worst imaginable symptom
Arm/Group | Placebo | Ropivacaine
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/33
Other Adverse Events (participants affected / at risk) | 20/38 | 18/33
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=38) | Ropivacaine (N=33)
Nausea (Gastrointestinal disorders) | 18 | 16
Pruritus (Skin and subcutaneous tissue disorders) | 20 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2018-04-26): https://cdn.clinicaltrials.gov/large-docs/44/NCT02829944/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2016-11-09): https://cdn.clinicaltrials.gov/large-docs/44/NCT02829944/Prot_SAP_001.pdf